CLINICAL TRIAL: NCT04427722
Title: A Multi-Centre Post Market Clinical Follow-Up Study of MPS-Flex® Total Knee Joint Prostheses in Total Knee Arthroplasty
Brief Title: PMCF Study of MPS-Flex® Knee System in TKA
Status: Suspended | Type: Observational
Why Stopped: No plan to extend CE mark
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSA2019-11K
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MPS-Flex Total Knee Joint Prostheses: Patients who have received MPS-Flex Total Knee Joint Prostheses for their primary TKA and meet the Patient Selection Criteria outlined in the study protocol.
  Interventions: Device: MPS-Flex Total Knee Joint Prostheses

INTERVENTIONS:
Device: MPS-Flex Total Knee Joint Prostheses — Patients who have received MPS-Flex Total Knee Joint Prostheses for their primary TKA and meet the Patient Selection Criteria outlined in the study protocol.

SUMMARY:
The objective of this study is to obtain implant survivorship and clinical outcomes data for the commercially available MPS-Flex® Total Knee Joint Prostheses used in primary total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
This is a retrospective and prospective, multi-centre, post-market clinical follow-up study involving orthopedic surgeons skilled in TKA and experienced implanting the devices included in this study. Patient demographic and operative information will be collected retrospectively. Postoperative clinical outcome, radiographic assessment and adverse events will be collected prospectively starting from the first year of postoperative follow up visit.

All study subjects have undergone routine preoperative clinical evaluations prior to their THA, and implanted MPS-Flex® Total Knee Joint Prostheses in accordance to indications and intended use, and appropriate surgical technique(s) will be invited to participate in the study at their first year of postoperative follow up visit, and sign ICF.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet the following criteria to be eligible for participation:

* Age 18 to 75 years old, inclusive.
* Had a primary unilateral or bilateral (simultaneous or staged)TKA based on physical exam and medical history, including diagnosis of severe knee pain and disability due to at least one of the following:

  1. Rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis.
  2. Collagen disorders and/or avascular necrosis of the femoral condyle.
  3. Post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy.
  4. Moderate valgus, varus, or flexion deformities.
* Had received MPS-Flex® Total Knee Joint Prostheses per the approved indications for use for the TKA.
* Willing and able to provide written informed consent by signing and dating the EC approved informed consent form.
* Willing and able to complete scheduled study procedures and follow-up evaluations.

Exclusion Criteria:

A patient must not meet the following criteria to be eligible for participation:

* The patient is:

  1. A prisoner
  2. Mentally incompetent or unable to understand what participation in the study entails
  3. A known alcohol or drug abuser
  4. Anticipated to be non-compliant
* Meet any of the following contraindications of the product.

  1. Had previous infection in the operative knee joint, and/or has systemic inflection that could affect prosthesis
  2. Insufficient bone stock of tibia or tibia surface
  3. Skeleton immaturity
  4. Neuropathic arthropathy
  5. Osteoporosis, muscle structure or neuromuscular lesions which affects lower limb function
  6. The affected joint occurs fusion in the satisfactory functional position and form stable,
  7. A history of rheumatoid arthritis with skin ulcers or recurrent skin damage
* Has a diagnosed systemic disease that could affect his/her safety or the study outcome.
* Known sensitivity or allergic reaction to one or more of the implanted materials.
* Known local bone tumors and/or cysts in the operative knee
* Known to be pregnant
* Body Mass Index (BMI) ≥ 40

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for primary statistical analysis will consist of patients who have already underwent their surgery with MPS-Flex® Total Knee Joint Prostheses for their primary TKA and satisfy eligibility criteria outlined in this section. In order to avoid potential selection bias, each investigator will offer study participation to each consecutive eligible patient presenting as a candidate for primary TKA using the MPS-Flex® Total Knee Joint Prostheses.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant survivorship based on revision | 10 years
  Implant survival will be summarized using a Kaplan-Meier method.

SECONDARY OUTCOMES:
Functional outcome based on Knee Society Score | 10 years
  The Knee Society Scoring System combines an objective physician-derived component with a subjective patient-derived component that evaluates pain relief, functional abilities, satisfaction, and fulfillment of expectations. It consists of four subscales: (1) Objective Knee Score (seven items; 100 points), (2) Satisfaction Score (five items; 40 points), (3) Expectation Score (three items; 15 points), and (4) Functional Activity Score (19 items; 100 points).
Quality of life based on EQ-5D questionnaire | 10 years
  EQ-5D is a standardized measure of health-related quality of life states consisting of 5 dimensions, namely mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L version was used in the study. Each dimension has 5 responses recording 5 levels of severity (no problems/slight problems/moderate problems/severe problems or extreme problems). The responses to the EQ-5D dimensions are used to obtain a single EQ-5D index value where 1 represents full health and 0 represents death. The questionnaire also includes a vertical, visual analogue scale (EQ VAS) for the respondents to record their self-rated health where the 2 extreme ends of the scale are labelled as 'Best imaginable health state' and 'Worst imaginable health state' respectively.
Safety assessment | 10 years
  Summarize the category, incidence and frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhong Guo, Professor, Principal Investigator — Jizhong Erengy Fengfeng Hospital
Locations (1):
- Jizhong Erengy Fengfeng Hospital, Handan, Hebei, China

IPD SHARING:
Plan to Share IPD: No